CLINICAL TRIAL: NCT02720978
Title: Tearing of Membranes Before Birth - a Comparison Between Two Ways of Induction of Labor Pitocin Opposite Prostaglandin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0073-15-TLV
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Fetus or Newborn or Maternal; Effects of Induction of Labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous oxytocin (Experimental): Women that arrive to women's ER and diagnosed with rupture of membranes in week 34+0 and onward, are not in active labor and with Bishop score lower than 7.
  Those who agreed to participate in the study after signing an informed consent form will undergo the following steps:
  1. Verification rupture of membranes and gestational age.
  2. Choosing the treatment group Intravenous oxytocin from red envelope, randomly.
  3. Collecting basic and obstetric data, laboratory results and physical examination, monitoring and sonar.
  4. Induction according to departmental protocol of each delivery way.
  5. Data collecting after the delivery.
  Interventions: Drug: Intravenous oxytocin
- vaginal prostaglandin (Experimental): Women that arrive to women's ER and diagnosed with rupture of membranes in week 34+0 and onward, are not in active labor and with Bishop score lower than 7.
  Those who agreed to participate in the study after signing an informed consent form will undergo the following steps:
  1. Verification rupture of membranes and gestational age.
  2. Choosing the treatment group vaginal prostaglandin from red envelope, randomly.
  3. Collecting basic and obstetric data, laboratory results and physical examination, monitoring and sonar.
  4. Induction according to departmental protocol of each delivery way.
  5. Data collecting after the delivery.
  Interventions: Drug: vaginal prostaglandin

INTERVENTIONS:
Drug: Intravenous oxytocin — Intravenous oxytocin chosen randomly. we will collect basic and obstetric data, laboratory results and physical examination, monitoring and sonar.
  Induction according to departmental protocol of each delivery way. Data collecting after the delivery.
  Arms: Intravenous oxytocin
Drug: vaginal prostaglandin — Vaginal prostaglandin chosen randomly. we will collect basic and obstetric data, laboratory results and physical examination, monitoring and sonar.
  Induction according to departmental protocol of each delivery way. Data collecting after the delivery.
  Arms: vaginal prostaglandin

SUMMARY:
Premature rupture of membranes (PROM) is a common occurrence that occurs in the incidence of 8-10% of births. Since the duration until delivery is important in avoiding the risk of complications, several studies have been performed in order to understand what is the preferred way to manage this condition of PROM in women that are not in active labor. In the largest random study that has been performed 20 years ago, there was found an advantage for labor induction with oxytocin over labor induction with Prostaglandin or waiting. However, the most important component - the BISHOP score, that affects the decision of the labor induction way, was not reported and was not taken into consideration.

DETAILED DESCRIPTION:
Premature rupture of membranes (PROM) is a common occurrence that occurs in the incidence of 8-10% of births. Since the duration until delivery is important in avoiding the risk of complications, several studies have been performed in order to understand what is the preferred way to manage this condition of PROM in women that are not in active labor. In the largest random study that has been performed 20 years ago, there was found an advantage for labor induction with oxytocin over labor induction with Prostaglandin or waiting. However, the most important component - the BISHOP score, that affects the decision of the labor induction way, was not reported and was not taken into consideration.

Therefore, the aim of the study is to compare randomly the perinatal outcomes in women with PROM and low BISHOP between women who undergo labor induction with Oxytocin and women who undergo labor induction with Prostaglandin E2.

ELIGIBILITY:
Inclusion Criteria:

1. rupture of membranes in BISHOP score lower than 7.
2. Pregnancy week 34+0 and onward.
3. Singleton pregnancy.
4. Verifying fetal monitoring.
5. Normal maternal temperature (lower than 37.8)
6. Without vaginal bleeding or suspected placental separation
7. Contractions in frequency of less than 3 in 10 minutes
8. Signed consent form.

Exclusion Criteria:

1. Multiple pregnancy.
2. Maternal age below 18 or over 42.
3. Active labor
4. Contractions in frequency of more than 3 in 10 minutes or cervical dilation ≥2 cm.
5. Lack of consent to participate in the study

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1200 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
The duration from the beginning of labor induction until delivery | 5 days

SECONDARY OUTCOMES:
Duration of labor induction from rupture of membranes until delivery. | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Maslovitz, MD, Principal Investigator — Tel Aviv Medical Center

IPD SHARING:
Plan to Share IPD: No